CLINICAL TRIAL: NCT06857825
Title: Effectiveness of Implementing an Infection Control Link Nurses Program to Improve Nurses' Compliance With Standard Precautions, Healthcare Professionals' Compliance With Hand Hygiene, and to Prevent Healthcare-Associated Infections: a Cluster Randomized Controlled Trial
Brief Title: Infection Control Link Nurses Program to Improve Compliance With Standard Precautions, Hand Hygiene, and Prevent Healthcare-Associated Infections
Acronym: INFECTION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Cardiologico Monzino (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CCM L2-284
Record Dates: First submitted 2025-02-27; First posted 2025-03-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Standard Precautions; Hand Hygiene Behavior; Healthcare Associated Infections
Keywords: Infection Control Link Nurse; Nursing; Hand Hygiene; Standard Precautions; Healthcare-associated infections
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Intervention Model Description: Cluster randomized control trial: all hospital wards and intensive care units of the promoting Center (i.e., n.8) will be divided in two parallel groups: 1) Intervention group (4 hospital units, implementation of one Infection Control Link Nurses per hospital unit); 2) Control group (4 hospital units, usual IPC practices) via cluster randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Infection Control Link Nurses (Experimental): In the Intervention group, in the 4 hospital medical-surgical wards and intensive care units randomized, will be implemented one infection control link nurse (ICLN) per hospital unit, for a total of 4 ICLNs They will receive ongoing education and they will be responsible for peer education about infection control practice, standard precaution measures, isolation measures, compliance with hand hygiene, promotion of evidence-based practice during patient care. They will act as a link between the IPC team and clinical practice, educating collegues and students on infection control guidelines
  Interventions: Behavioral: Implementation of Infection Control Link Nurses (ICLNs)
- Control group (No Intervention): In the Control group, 4 hospital medical-surgical wards and intensive care units will continue their normal practice, following usual IPC measures

INTERVENTIONS:
Behavioral: Implementation of Infection Control Link Nurses (ICLNs) — Infection Control Link Nurses (ICLNs) are clinical nurses, working in direct nursing care, with an interest and expertise on infection control practice. They work with constant and direct support by the IPC hospital team, and they are required to follow a training course with numerous scheduled meetings about IPC-related issues.
  They will be selected via spontaneous application or identified by their Head Nurses. All ICLNs activities are to be completed during working hours, they still maintain their clinical nursing role, but in addition they implement and translate IPC-measures into clinical practice by observing, monitoring and analyzing data on compliance with hand hygiene, compliance with standard and isolation precautions, healthcare-associated infections and other IPC-related issues
  Arms: Infection Control Link Nurses

SUMMARY:
The goal of this clinical trial is to learn if Infection Control Link Nurses (i.e., clinical nurses providing direct patient care with an interest and expertise in infection control practices) are effective in improving nurses' compliance with standard precaution measures, healthcare professional's compliance with hand hygiene practices and in reducing healthcare-associated infections. The main questions it aims to answer are:

* Are Infection Control Link Nurses effective in improving nurses' compliance with standard precautions?
* Are Infection Control Link Nurses effective in improving healthcare professionals' compliance with hand hygiene practices?
* Are Infection Control Link Nurses effective in improving alcohol-based hand rub consumption?
* Are Infection Control Link Nurses effective in reducing healthcare-associated infections? In this study, a total of 8 hospital units will be randomized in two groups: 1) Intervention group, where in 4 hospital units will be selected and trained 4 Infection Control Link Nurses; and 2) Control group, where in 4 hospital units will continue usual IPC practice.

Training of Infection Control Link Nurses will be 12 months-long, with regular monthly scheduled meetings.

Researchers will compare Intervention group with the Control group to see if nurses' compliance with standard precautions and healthcare professionals' compliance with hand hygiene will improve in the Intervention group, and if overall healthcare-associated infection incidence will decrease.

Participants will be nurses working full time in the selected hospital units, for a total of 100 nurses. They will sign an Informed Consent form and they will fill out a validated instrument named "Compliance with Standard Precautions Scale-Italian Version", to measure their adherence to standard precautions measures (i.e., use of protective device, disposal of sharp, disposal of waste etc). Concurrently, evaluation of healthcare professionals' compliance with hand hygiene will be done via direct observation, following World Health Organization's Technical Manual, by hospital staff who did not participate in the conception and design of the study. Lastly, data regarding alcohol-based hand rub consumption and healthcare-associated infections will be collected by experienced personnel who routinely perform these activities. The study will last 12 months, data collection will be carried out at baseline (pre-implementation of infection control link nurses) and after 12 months (after infection control link nurses implementation).

DETAILED DESCRIPTION:
In this cluster RCT, all medical-surgical wards and ICUs of the Center where the study will be conducted, will be selected. Subsequently, cluster randomization will divide those hospital units in two arms: (1) Intervention group - 1 ICLN per ward/ICU will be identified and formed; (2) Control group - wards and ICU that will continue standard IPC practice.

Assessment, data collection, and intervention will be administered within the hospital facility. Since this hospital comprises in total 6 medical-surgical wards and 2 ICUs, each study group (i.e., Intervention group and Control group) will comprise 4 hospital units.

Data will be collected in presence at baseline (T0 - before ICLNs' implementation) and after 12 months (T1).

* Primary endpoint will be nurses' compliance with standard precautions, using a validated instrument ("Compliance with Standard Precaution Scale-Italian version; CSPS-It)
* Secondary outcomes (i.e., healthcare professionals' hand hygiene compliance, healthcare professionals' alchol-based hand rub consumption and healthcare-associated infections incidence rate) will be evaluated for all healthcare professionals working in the promoting center.

Signing of Informed Consent will only be required by nursing staff who fill-out the CSPS-It, whereas all other data collected (hand hygiene compliance, alchol-based hand rub consumption consumption and HAIs incidence) are part of usual intra-hospital surveillance practices and do not involve the collection of any personal data.

For this reason, nurses working in the selected units will be asked to participate in the study, and they will be asked to sign an Informed Consent form and will be consecutively enrolled until the sample size is reached (i.e., 100 nurses).

After cluster randomization is performed, recruitment of potential participants will begin. 4 ICLNs will be selected and every clinical nurse working full-time in the selected hospital units will be asked to participate in the present RCT. After signing the Informed Consent, baseline data collection will begin.

At baseline (T0) socio-demographic data and job-related informations (e.g., time in years of clinical experience as a nurse, study degree) will be collected. Afterward, participants will be asked to fill out a validated instrument aiming to measure compliance with standard precautions (i.e., CSPS-it). Sample size is composed only by nurses because CSPS-It is validated only for registered nurses and nursing students.

Concurrently, data regarding healthcare professionals' (i.e., doctors, nurses, support personnel, technicians) compliance with hand hygiene (HH), Alcohol-Based Hand Rub (ABHR) consumption, and Healthcare-Associated Infections (HAIs)' incidence rate will be collected.

During the 12-month ICLNs implementation program, ICLNs will be continuously supported in their activities by hospital management and by their colleagues, and they will be asked to participate in monthly educational meetings covering core elements on HAIs prevention and control, standard and isolation precaution measures, and hand hygiene paired with flexible times useful for ICLNs to create debates, reflect on barriers, and analyze situations together.

After 12 months (T1), the same data collection at baseline (T0) will be performed (i.e., CSPS-it, HH compliance, ABHR consumption, HAIs' incidence rate).

Data collection will be carried out by research assistants trained to the present protocol, HH compliance direct observations will be performed by hospital personnel not involved in this RCT, data related to AHRB consumption and HAIs rate will be collected by trained personnel working in the hospital facility.

To ensure privacy, data at baseline and follow-up will be collected, analyzed and presented exclusively in aggregate form (i.e., for the intervention group and control group).

ELIGIBILITY:
Inclusion Criteria:

* Nursing staff working full time in the hospital wards and intensive care units partecipating in the study

Exclusion Criteria:

* Nurses unavailable to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Nurses' compliance with standard precautions | Data will be collected at enrollment (baseline), and at the end of study (12 months after baseline)
  Standard Precautions are measure that healthcare professionals need to apply into practice with dual aim: to protect themselves from contamination during direct patient care, and to prevent/reduce healthcare-associated infections in patients. It will be measured via the Compliance with Standard Precaution Scale, Italian version (CSPS-It). Written approval and permission to use the scale have been obtained both by the original author and by the author of the Italian-validated version. CSPS-It is a 20-item instrument, validated for registered nurses and nursing students, aiming to assess nursing staff's compliance with standard precautions measures (e.g., use of protective device, disposal of sharp, disposal of waste). It comprises 20 items, both positively and negatively worded, answerable with a 4-point Likert scale ranging from 1 ("never") to 4 ("always"). Scoring ranges between 0 and 20, with higher scores reflecting better compliance with standard precautions

SECONDARY OUTCOMES:
Healthcare professionals' compliance with hand hygiene | Data will be collected at enrollment (baseline), and at the end of study (12 months after baseline)
  Healthcare professionals' hand hygiene compliance will be evaluated via direct observation, following the World Health Organization - Hand Hygiene Technical Reference Manual. This Manual explains in detail how an observer should conduct the evaluation, following the 5 moments for hand hygiene (1. Before touching a patient; 2. Before clean/aseptic procedure; 3. After body fluid exposure risk; 4. After touching a patient; 5. After touching patient surroundings) defined by WHO to clean healthcare professionals' hands with soap and water or AHRB. WHO Technical Reference Manual contains a specific part (i.e., Part III - Observing hand hygiene practices) that guides step by step direct observations of HH. Calculation % of HH compliance of the observed staff is based on the following formula: Compliance (%)= (Performed actions/Opportunities) x 100.
Alchol-Based Hand Rub (ABHR) consumption | Data will be collected at enrollment (baseline), and at the end of study (12 months after baseline)
  Alchol-based hand rub (ABHR) consumption is a proxy measure of hand hygiene. It involves measuring the quantity of hydro-alcoholic hand sanitizing solution used by healthcare professionals in a set period of time, through consumption flows. ABHR consumption will be analyzed via the following equation, proposed by WHO: (ABHR consumption)/(1000 patient-days). WHO proposes a rate of ABHR consumption >=20 Liters/1000 patient-days as the desirable standard.
Incidence of Healthcare-Associated Infections (HAIs) | Data will be collected at enrollment (baseline), and at the end of study (12 months after baseline)
  Incidence of the following Healthcare-Associated Infections (HAIs) will be calculated: catheterization-associated urinary tract infections (CAUTIs), mechanical ventilation-associated pneumonia (VAPs), surgical site infections (SSIs) and bloodstream infections (BSIs). The incidence rate of VAP, CAUTI, SSI, and BSI will be calculated as per the usual reporting of positive culture specimens by the CCM Medical Laboratory. All first positive culture samples associated with a specific hospital unit will be considered. Individual cases will then be analyzed, by experienced personnel who routinely perform these activities, based on the Atlanta Center of Disease Control Guidelines, identifying hospital HAIs. Incidence of each HAI (i.e., VAP, CAUTI, SSI, BSI) will be calculated using the following equation:
  Incidence rate= (Number of first positive cultures per patient / Number of unit's admissions) x 1000 patient-days

CONTACTS AND LOCATIONS:
Overall Officials: Miriana D'Andrea, Master of Science in Nursing, Principal Investigator — Centro Cardiologico Monzino, IRCCS, 20138 Milan, Italy.
Locations (1):
- Centro Cardiologico Monzino, IRCCS, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ojanpera H, Kanste OI, Syrjala H. Hand-hygiene compliance by hospital staff and incidence of health-care-associated infections, Finland. Bull World Health Organ. 2020 Jul 1;98(7):475-483. doi: 10.2471/BLT.19.247494. Epub 2020 May 26. PMID 32742033
- [Background] Dekker M, Jongerden IP, Caris MG, de Bruijne MC, Vandenbroucke-Grauls CMJE, van Mansfeld R. Evaluation of an infection control link nurse program: an analysis using the RE-AIM framework. BMC Health Serv Res. 2023 Feb 9;23(1):140. doi: 10.1186/s12913-023-09111-5. PMID 36759832
- [Background] Ghorbanmovahhed S, Shahbazi S, Gilani N, Ostadi A, Shabanloei R, Gholizadeh L. Effectiveness of implementing of an infection control link nurse program to improve compliance with standard precautions and hand hygiene among nurses: a quasi-experimental study. BMC Med Educ. 2023 Apr 19;23(1):265. doi: 10.1186/s12909-023-04208-1. PMID 37076871
- [Background] Sopirala MM, Yahle-Dunbar L, Smyer J, Wellington L, Dickman J, Zikri N, Martin J, Kulich P, Taylor D, Mekhjian H, Nash M, Mansfield J, Pancholi P, Howard M, Chase L, Brown S, Kipp K, Lefeld K, Myers A, Pan X, Mangino JE. Infection control link nurse program: an interdisciplinary approach in targeting health care-acquired infection. Am J Infect Control. 2014 Apr;42(4):353-9. doi: 10.1016/j.ajic.2013.10.007. Epub 2014 Feb 16. PMID 24548456
- [Background] Donati D, Miccoli GA, Cianfrocca C, Di Stasio E, De Marinis MG, Tartaglini D. Effectiveness of implementing link nurses and audits and feedback to improve nurses' compliance with standard precautions: A cluster randomized controlled trial. Am J Infect Control. 2020 Oct;48(10):1204-1210. doi: 10.1016/j.ajic.2020.01.017. Epub 2020 Mar 13. PMID 32178856
- [Background] Dekker M, van Mansfeld R, Vandenbroucke-Grauls C, de Bruijne M, Jongerden I. Infection control link nurse programs in Dutch acute care hospitals; a mixed-methods study. Antimicrob Resist Infect Control. 2020 Feb 27;9(1):42. doi: 10.1186/s13756-020-0704-2. PMID 32106884
- [Background] Cusumaro C, Ocagli H. [The Healthcare-associated infections (HAIs) and infection Control link nurse as a strategy to face them: review of literature]. Prof Inferm. 2021 Jul-Sep;74(3):153-160. doi: 10.7429/pi.2021.742153. Italian. PMID 35084158
- [Background] Dekker M, van Mansfeld R, Vandenbroucke-Grauls CM, Lauret TE, Schutijser BC, de Bruijne MC, Jongerden IP. Role perception of infection control link nurses; a multi-centre qualitative study. J Infect Prev. 2022 May;23(3):93-100. doi: 10.1177/17571774211066786. Epub 2022 Feb 18. PMID 35495104
- [Background] Peter D, Meng M, Kugler C, Mattner F. Strategies to promote infection prevention and control in acute care hospitals with the help of infection control link nurses: A systematic literature review. Am J Infect Control. 2018 Feb;46(2):207-216. doi: 10.1016/j.ajic.2017.07.031. PMID 29413157
- [Background] Dawson SJ. The role of the infection control link nurse. J Hosp Infect. 2003 Aug;54(4):251-7; quiz 320. doi: 10.1016/s0195-6701(03)00131-2. PMID 12919754
- [Background] Dekker M, Jongerden IP, van Mansfeld R, Ket JCF, van der Werff SD, Vandenbroucke-Grauls CMJE, de Bruijne MC. Infection control link nurses in acute care hospitals: a scoping review. Antimicrob Resist Infect Control. 2019 Jan 28;8:20. doi: 10.1186/s13756-019-0476-8. eCollection 2019. PMID 30705754
- [Background] Dekker M, Jongerden IP, van Mansfeld R. Implementation of infection prevention in intensive and critical care: What an infection control link nurse can contribute. Intensive Crit Care Nurs. 2024 Aug;83:103705. doi: 10.1016/j.iccn.2024.103705. Epub 2024 Apr 16. No abstract available. PMID 38631276
- [Background] Brusaferro S, Arnoldo L, Cattani G, Fabbro E, Cookson B, Gallagher R, Hartemann P, Holt J, Kalenic S, Popp W, Privitera G, Prikazsky V, Velasco C, Suetens C, Varela Santos C. Harmonizing and supporting infection control training in Europe. J Hosp Infect. 2015 Apr;89(4):351-6. doi: 10.1016/j.jhin.2014.12.005. Epub 2015 Jan 7. PMID 25777079
- See also: Royal College of Nursing. The Role of the Link Nurse in Infection Prevention and Control (IPC): developing a link nurse framework. RCN — https://www.rcn.org.uk/Professional-Development/publications/rcn-role-of-the-link-nurse-in-infection-prevention-and-control-uk-pub-009595
- See also: European Centre for Disease Prevention and Control. Point prevalence survey of healthcare-associated infections and antimicrobial use in European acute care hospitals, 2022-2023. — https://data.europa.eu/doi/10.2900/88011